CLINICAL TRIAL: NCT04191733
Title: Prospective, Randomized, Multi-center Post-Market Study of Anterior Advantage Surgical Approach in Total Hip Arthroplasty With and Without the KINCISE™ Surgical Automated System.
Brief Title: Anterior Advantage With KINCISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study early. Data collection was sufficient to adequately assess primary endpoint.
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSJ_2019_03
Record Dates: First submitted 2019-10-28; First posted 2019-12-10 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: 1:1 Block Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anterior Approach with KINCISE (Experimental): Anterior Approach THA using KINCISE(TM) Surgical Automated System
  Interventions: Device: KINCISE(TM) Surgical Automated System
- Anterior Approach without KINCISE (Active Comparator): Anterior Approach THA with a mallet (without KINCISE)
  Interventions: Device: KINCISE(TM) Surgical Automated System

INTERVENTIONS:
Device: KINCISE(TM) Surgical Automated System — Uncemented Total Hip Arthroplasty via Anterior Approach with and without the KINCISE(TM) Surgical Automated System

SUMMARY:
This is a post-market prospective, 1:1 randomized, multicenter non-inferiority study to compare the femoral broaching time for THA with the Anterior Advantage approach with KINCISE vs. without KINCISE. Follow-up will continue through 24 weeks post-op.

DETAILED DESCRIPTION:
The primary endpoint is femoral broaching time (in minutes), which is collected intraoperatively. The primary objective is to demonstrate that femoral broaching time with KINCISE is non-inferior to femoral broaching time with manual instruments (not using KINCISE) when used in THA with Anterior Advantage.

Note: If non-inferiority is successfully demonstrated, then the study will be deemed to be successful, and a test for superiority of femoral broaching time will be conducted.

If the primary endpoint analysis successfully demonstrates non-inferiority of femoral broaching time, then the following three secondary objectives will be assessed with formal hypotheses, in order, under a gatekeeping strategy:

* Non-inferiority of skin-to-skin OR time when KINCISE is used vs. when KINCISE is not used.
* Non-inferiority of the percent of subjects with optimal acetabular cup abduction angle when KINCISE is used vs. when KINCISE is not used.
* Non-inferiority of the percent of subjects with optimal acetabular cup version angle when KINCISE is used vs. when KINCISE is not used.

In addition, the following secondary endpoints do not have prospectively planned hypotheses; these will be summarized for both treatment groups:

* Harris Hip Score (HHS) and HHS change from preoperative baseline
* Forgotten Joint Score (FJS) and FJS change from 6-week postoperative baseline
* EQ-5D-5L and changes in these assessments from preoperative baseline
* Pain (Groin, Thigh, and Buttock)
* Patient Satisfaction
* Post-op time when functional activities can be accomplished (return to work, self-care, etc.)
* Radiographic Outcomes (based upon AP Hip, AP Pelvis, and Lateral)
* Length of hospital stay after index THA
* Re-hospitalizations during the study (including a specific summary of re-hospitalizations within 90 days)
* Narcotic drug usage throughout the study (participant reported)
* Complications (including a specific summary of complications within 90 days post-surgery)

ELIGIBILITY:
Inclusion Criteria:

1. The patient is undergoing a standard of care primary cementless hip replacement with the Pinnacle cup and a Corail or Actis stem via the Anterior Advantage approach. All devices are to be used according to the approved indications.
2. Individuals who are able to speak, read, and comprehend the Institutional Review Board approved Informed Consent Document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes.
3. Individuals who are willing and able to complete follow-up visits and questionnaires as specified by the study protocol.
4. Individuals who are not bedridden per the discretion of the investigator (The intent of "not bedridden" means a permanent situation, not a temporary situation as in a hip fracture or trauma case).
5. Individuals who are a minimum age of 21 years at the time of consent.

Exclusion Criteria:

1. Active local or systemic infection.
2. Loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
3. Poor bone quality, such as osteoporosis, where, in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
4. Charcot's or Paget's disease.
5. The Subject is a woman who is pregnant or lactating.
6. Subject had a contralateral amputation.
7. Previous partial hip replacement in affected hip.
8. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
9. Contralateral hip was replaced less than 3 months prior to surgery date, contralateral hip is already enrolled in the study, or simultaneous or staged hip replacement is planned
10. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
11. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
12. Subject has a medical condition with less than 2 years of life expectancy.
13. Subject, in the opinion of the Investigator, is a drug or alcohol abuser or has a physical or psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - The Orthopedic Specialty Center of Northern California, Roseville, California
  - Colorado Joint Replacement, Denver, Colorado
  - Capital Region Orthopaedic Group, Albany, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolina Orthopaedic & Sports Medicine, Gastonia, North Carolina
  - Southern Joint Replacement Institute, Nashville, Tennessee
  - Texas Institute for Hip and Knee Surgery, Austin, Texas
  - W.B. Carrell Memorial Clinic, Dallas, Texas
  - North Texas Medical Research Institute, Dallas, Texas
  - Jordan-Young Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu/
URL: http://yoda.yale.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 250 participants were enrolled in this study, out of which 7 participants withdrew study before assignment to any treatment. Hence, only 243 participants were included in the analysis.
Groups:
- Arm 1: KINCISE: Participants indicated to receive primary uncemented total hip arthroplasty (THA) underwent Anterior Advantage approach in THA using KINCISE surgical automated system.
- Arm 2: MALLET: Participants indicated to receive primary uncemented THA underwent Anterior Advantage approach in THA using MALLET (a surgical hammer like instrument, without KINCISE surgical automated system).
Period: Overall Study
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Started (Enrolled participants) | 122 | 121
Enrolled But Not Treated | 5 | 10
Safety Population (The safety population set consisted of all enrolled participants who signed the informed consent document and attempted treatment according to the actual treatment received.) | 117 | 111
Completed | 101 | 95
Not Completed | 21 | 26
Not completed — Withdrawn due to study closure | 13 | 14
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 5 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population set consisted of all enrolled participants who signed the informed consent document and attempted treatment according to the actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET | Total
Number analyzed (Participants) | 117 | 111 | 228
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.65) | 64.5 (9.42) | 64.4 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 55 | 49 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 88 | 82 | 170
  Unknown or Not Reported | 29 | 26 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 101 | 89 | 190
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Femoral Broach Time
Description: Mean femoral broach time (in minutes) was collected intraoperatively and begun at the time the box osteotome first enters the femoral canal and ended with seating of the final broach trial within the femoral canal.
Time Frame: Day 0 (operative day)
Population: Per protocol population set consisted of all enrolled participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, and who did not have any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 107 | 109
Minutes | 5.8 (4.01) | 8.1 (6.06)
Statistical Analysis 1: Comparison: Arm 1: KINCISE vs Arm 2: MALLET; Test type: Non-Inferiority — The non-inferiority analysis was demonstrated when the 1-sided upper 95% confidence interval (CI) limit was less than 1.25; p < 0.0001, t-test, 1 sided — one-sided p-value

2. Secondary Outcome: Skin-to-skin Time
Description: Skin-to-skin is the time (in minutes) duration of the surgery procedure.
Time Frame: Day 0 (operative day)
Population: Per protocol population set consisted of all enrolled participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, and who did not have any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 109 | 109
Minutes | 71.0 (18.15) | 70.2 (15.61)
Statistical Analysis 1: Comparison: Arm 1: KINCISE vs Arm 2: MALLET; A gatekeeping strategy was used to control family-wise type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The testing sequence continued only when previous endpoint was statistically significant with a 1-sided alpha of 0.05; Test type: Non-Inferiority — 1-sided test with 5% alpha was used to demonstrate non-inferiority with greater than 99% power. The non-inferiority margin was 3.75 minutes; p = 0.1004, t-test, 1 sided

3. Secondary Outcome: Number of Participants With Optimal Acetabular Cup Abduction Angle at Week 6
Description: Number of participants with optimal acetabular cup (a socket of the hip joint) abduction angle (movement of the leg away from the midline of the body) within +/- 10 degree of plan at Week 6 was reported.
Time Frame: At Week 6 (post operative)
Population: Per protocol population set consisted of all enrolled participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, and who did not had any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Participants | 98 | 95

4. Secondary Outcome: Number of Participants With Optimal Acetabular Cup Version Angle at Week 6
Description: Number of participants with optimal acetabular cup (a socket of the hip joint) version angle (rotation of leg in hip joint) within +/- 10 degrees of plan at Week 6 was reported.
Time Frame: At Week 6 (post operative)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 101 | 94
Participants | 93 | 88

5. Secondary Outcome: Change From Pre-operative Baseline in Harris Hip Score (HHS) at Weeks 6 and 24
Description: The HHS was developed for the assessment of the results of hip surgery. HHS was intended to evaluate various hip disabilities and methods of treatment in an adult population. It consisted of 10 items covering four domains: pain (1 item, 0-44 points), function ( 7 items [limb, support, distance walked, stairs, socks/shoes, sitting and public transportation], 0-47 points), deformity (1 item, 4 points) and range of hip motion (1 items, 5 points). HHS total score was the sum of 10 items scores and ranged from 0 (worse disability) to 100 (less disability). The higher score indicated better outcome for the participant. The scores were interpreted as follows: < 70 = poor, 70-79 = fair, 80-89 = good and 90-100 = excellent. Day 0 was the operative day.
Time Frame: Pre-operative baseline (6 months before operative day), 6 weeks and 24 weeks post-operative
Population: Per protocol population set consisted of all enrolled participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, who did not had any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data. 'N'(number of participants analyzed)=who were evaluable for this outcome measure, 'n'(number analyzed)=participant who were evaluated at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 100 | 98
Units on a scale
  Week 6 | 29.0 (18.32) | 27.3 (18.95)
  Week 24: number analyzed (Participants) | 94 | 92
  Week 24 | 38.7 (14.43) | 41.0 (14.93)

6. Secondary Outcome: Change From 6-week Post-surgery in Forgotten Joint Score (FJS-12) at Week 24
Description: The FJS was a 12 question form that asks the participants their level of awareness of their artificial joint in 12 scenarios commonly encountered in daily life. Response to each question was individually scored (0 to 4, where 0=never, 1=almost never, 2=seldom, 3=sometimes and 4=mostly) and summed to create a raw composite score that was normalized to a range of 0 to 100 with a higher score indicating a better outcome (high degree of forgetting the artificial joint in everyday life).
Time Frame: 6-week post-operative to 24 weeks post-operatively
Population: Per protocol population set consisted of all participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, who did not had any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data. Here, 'N' (number of participants analyzed)=who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 87 | 84
Units on a scale | 25.3 (27.68) | 22.2 (26.40)

7. Secondary Outcome: Change From Pre-operative Baseline in European Quality of Life (EuroQol)-5 Dimension-5 Level (EQ-5D-5L) Heath State Index Total Score at Weeks 6 and 24
Description: EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses to 5 EQ-5D-5L dimensions were scored using a utility-weighted algorithm to derive an EQ-5D-5L health status index score between 0 (death) to 100 (full health). Higher score indicated better QoL.
Time Frame: Pre-operative baseline (6 months before operative day), 6 weeks and 24 weeks post-operative
Population: Per protocol population set consisted of all participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, who did not had any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data. Here, 'N'(number of participants analyzed)=who were evaluable for this outcome measure, 'n'(number analyzed)=participant who were evaluated at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 100 | 97
Units on a scale
  Week 6 | 0.18 (0.164) | 0.16 (0.187)
  Week 24: number analyzed (Participants) | 94 | 91
  Week 24 | 0.25 (0.162) | 0.28 (0.173)

8. Secondary Outcome: Change From Pre-operative Baseline in EQ-5D-5L Visual Analog Scale (VAS) Total Score at Weeks 6 and 24
Description: EQ-5D-5L was a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a vertical line VAS with scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). A higher score indicates better health and positive changes from baseline indicate improvement of health status.
Time Frame: Pre-operative baseline (6 months before operative day), 6 weeks and 24 weeks post-operative
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 100 | 98
Units on a scale
  Week 6 | 12.3 (16.52) | 10.0 (16.52)
  Week 24: number analyzed (Participants) | 95 | 92
  Week 24 | 12.8 (15.26) | 11.9 (17.97)

9. Secondary Outcome: Number of Participants With Pain (Groin, and Buttock) at Weeks 6 and 24
Description: Number of participants with pain (Groin, and Buttock) at Weeks 6 and 24 was reported. Participant's groin pain and buttock pain was reported either as none, mild, moderate, or severe.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 102 | 98
Participants
  Week 6: Groin pain: None | 57 | 60
  Week 6: Groin pain: Mild | 38 | 27
  Week 6: Groin pain: Moderate | 6 | 11
  Week 6: Groin pain: Severe | 0 | 0
  Week 6: Groin pain: Missing | 1 | 0
  Week 24: Groin pain: number analyzed (Participants) | 95 | 93
  Week 24: Groin pain: None | 78 | 72
  Week 24: Groin pain: Mild | 15 | 18
  Week 24: Groin pain: Moderate | 1 | 2
  Week 24: Groin pain: Severe | 1 | 1
  Week 24: Groin pain: Missing | 0 | 0
  Week 6: Buttock pain: None | 66 | 61
  Week 6: Buttock pain: Mild | 31 | 30
  Week 6: Buttock pain: Moderate | 5 | 6
  Week 6: Buttock pain: Severe | 0 | 1
  Week 6: Buttock pain: Missing | 0 | 0
  Week 24: Buttock pain: number analyzed (Participants) | 95 | 93
  Week 24: Buttock pain: None | 81 | 80
  Week 24: Buttock pain: Mild | 11 | 11
  Week 24: Buttock pain: Moderate | 2 | 2
  Week 24: Buttock pain: Severe | 1 | 0
  Week 24: Buttock pain: Missing | 0 | 0

10. Secondary Outcome: Number of Participants With Post-operative Satisfaction With the Procedure at Weeks 6 and 24
Description: Number of participants with post-operative satisfaction with the procedure at Weeks 6 and 24 was reported. Participants were asked a question that "How satisfied do you anticipate you will be with this procedure?" and participant responded on a 5-point scale (1=extremely satisfied, 2=very satisfied, 3=moderately satisfied, 4=slightly satisfied, 5=not at all satisfied). Higher score indicated low post-operative satisfaction.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 102 | 98
Participants
  Week 6: Extremely satisfied | 80 | 66
  Week 6: Very satisfied | 15 | 23
  Week 6: Moderately satisfied | 5 | 6
  Week 6: Slightly satisfied | 0 | 2
  Week 6: Not at all satisfied | 1 | 0
  Week 6: Missing | 1 | 1
  Week 24: number analyzed (Participants) | 95 | 93
  Week 24: Extremely satisfied | 78 | 77
  Week 24: Very satisfied | 13 | 12
  Week 24: Moderately satisfied | 2 | 2
  Week 24: Slightly satisfied | 1 | 0
  Week 24: Not at all satisfied | 1 | 2
  Week 24: Missing | 0 | 0

11. Secondary Outcome: Number of Participants With Post-operative Functional Recovery at Week 6
Description: Participants were asked the following questions: "Can you walk without an aid?", "Do you drive?", "Can you perform basic activities of daily living without assistance?", "Can you perform light household duties?", "Can you perform moderate to heavy household duties?", "Can you go up and down a flight of stairs using a handrail?", "Can you put on socks/stockings without someone's assistance?", "Can you bend down to pick up an object on the floor?", "Can you stand up from a chair without assistance?", "Can you participate in leisure recreational activities?", "Do you work?" and "When were you first able to accomplish the primary goal you identified after surgery?". Participants were asked to respond either as "yes" or "No, because of study hip". Number of participants who reported response as "yes" at Week 6 were reported in this outcome measure.
Time Frame: Week 6 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 106 | 107
Participants
  Can you walk without an aid?: number analyzed (Participants) | 102 | 101
  Can you walk without an aid? | 96 | 95
  Do you drive?: number analyzed (Participants) | 106 | 97
  Do you drive? | 98 | 93
  Can you perform basic activities of daily living without assistance?: number analyzed (Participants) | 106 | 105
  Can you perform basic activities of daily living without assistance? | 104 | 103
  Can you perform light household duties?: number analyzed (Participants) | 103 | 102
  Can you perform light household duties? | 100 | 99
  Can you perform moderate to heavy household duties?: number analyzed (Participants) | 95 | 91
  Can you perform moderate to heavy household duties? | 75 | 68
  Can you go up and down a flight of stairs using a handrail?: number analyzed (Participants) | 100 | 100
  Can you go up and down a flight of stairs using a handrail? | 96 | 96
  Can you put on socks/stockings without someone's assistance?: number analyzed (Participants) | 105 | 102
  Can you put on socks/stockings without someone's assistance? | 94 | 90
  Can you bend down to pick up an object on the floor?: number analyzed (Participants) | 103 | 105
  Can you bend down to pick up an object on the floor? | 98 | 98
  Can you stand up from a chair without assistance?: number analyzed (Participants) | 103 | 107
  Can you stand up from a chair without assistance? | 102 | 104
  Can you participate in leisure recreational activities?: number analyzed (Participants) | 90 | 86
  Can you participate in leisure recreational activities? | 65 | 52
  Do you work?: number analyzed (Participants) | 51 | 48
  Do you work? | 46 | 37
  When were you first able to accomplish primary goal you identified after surgery?: number analyzed (Participants) | 106 | 104
  When were you first able to accomplish primary goal you identified after surgery? | 62 | 63

12. Secondary Outcome: Number of Participants With Radiographic Outcomes: Assessed on Acetabular Cup, Femoral Stem, Calcar Resorption and Calcar Fractur
Description: Number of participants with radiographic outcomes (acetabular cup migration, acetabular cup radiolucency, acetabular cup progressive radiolucency, acetabular cup osteolysis, acetabular cup sclerotic lines, acetabular cup porous coating integrity, femoral stem subsidence, femoral stem radiolucency, femoral stem osteolysis, calcar resorption, calcar fracture, femoral stem tilt and femoral stem porous coating integrity) were reported. In this outcome measure, only those timepoints in which participants had data were reported. In this outcome measure, each radiographic outcome assessment was reported either as present or absent in the analyzed participants.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Participants
  Week 24: Acetabular Cup Migration: Present: number analyzed (Participants) | 93 | 92
  Week 24: Acetabular Cup Migration: Present | 0 | 0
  Week 24: Acetabular Cup Migration: Absent: number analyzed (Participants) | 93 | 92
  Week 24: Acetabular Cup Migration: Absent | 93 | 92
  Week 6: Acetabular Cup Radiolucency: Present | 0 | 0
  Week 6: Acetabular Cup Radiolucency: Absent | 103 | 99
  Week 24: Acetabular Cup Radiolucency: Present: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Radiolucency: Present | 0 | 0
  Week 24: Acetabular Cup Radiolucency: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Radiolucency: Absent | 95 | 93
  Week 24: Acetabular Cup Progressive Radiolucency: Present: number analyzed (Participants) | 91 | 88
  Week 24: Acetabular Cup Progressive Radiolucency: Present | 0 | 0
  Week 24: Acetabular Cup Progressive Radiolucency: Absent: number analyzed (Participants) | 91 | 88
  Week 24: Acetabular Cup Progressive Radiolucency: Absent | 91 | 88
  Week 24: Acetabular Cup Osteolysis: Present: number analyzed (Participants) | 93 | 92
  Week 24: Acetabular Cup Osteolysis: Present | 0 | 0
  Week 24: Acetabular Cup Osteolysis: Absent: number analyzed (Participants) | 93 | 92
  Week 24: Acetabular Cup Osteolysis: Absent | 93 | 92
  Week 6: Acetabular Cup Sclerotic Lines: Present | 0 | 0
  Week 6: Acetabular Cup Sclerotic Lines: Absent | 103 | 99
  Week 24: Acetabular Cup Sclerotic Lines: Present: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Sclerotic Lines: Present | 0 | 0
  Week 24: Acetabular Cup Sclerotic Lines: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Sclerotic Lines: Absent | 95 | 93
  Week 6: Acetabular Cup Porous Coating Integrity: Present | 0 | 0
  Week 6: Acetabular Cup Porous Coating Integrity: Absent | 103 | 99
  Week 24: Acetabular Cup Porous Coating Integrity: Present: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Porous Coating Integrity: Present | 0 | 0
  Week 24: Acetabular Cup Porous Coating Integrity: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Porous Coating Integrity: Absent | 95 | 93
  Week 24: Femoral Stem Subsidence: Present: number analyzed (Participants) | 93 | 92
  Week 24: Femoral Stem Subsidence: Present | 0 | 0
  Week 24: Femoral Stem Subsidence: Absent: number analyzed (Participants) | 93 | 92
  Week 24: Femoral Stem Subsidence: Absent | 93 | 92
  Week 6: Femoral Stem Radiolucency: Present | 0 | 0
  Week 6: Femoral Stem Radiolucency: Absent | 103 | 99
  Week 24: Femoral Stem Radiolucency: Present: number analyzed (Participants) | 95 | 93
  Week 24: Femoral Stem Radiolucency: Present | 0 | 1
  Week 24: Femoral Stem Radiolucency: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Femoral Stem Radiolucency: Absent | 95 | 92
  Week 24: Femoral Stem Osteolysis: Present: number analyzed (Participants) | 93 | 92
  Week 24: Femoral Stem Osteolysis: Present | 1 | 0
  Week 24: Femoral Stem Osteolysis: Absent: number analyzed (Participants) | 93 | 92
  Week 24: Femoral Stem Osteolysis: Absent | 92 | 92
  Week 6: Calcar Resorption: Present | 0 | 0
  Week 6: Calcar Resorption: Absent | 103 | 99
  Week 24: Calcar Resorption: Present: number analyzed (Participants) | 95 | 93
  Week 24: Calcar Resorption: Present | 1 | 2
  Week 24: Calcar Resorption: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Calcar Resorption: Absent | 94 | 91
  Week 6: Calcar Fracture: Present | 0 | 0
  Week 6: Calcar Fracture: Absent | 103 | 99
  Week 24: Calcar Fracture: Present: number analyzed (Participants) | 95 | 93
  Week 24: Calcar Fracture: Present | 0 | 0
  Week 24: Calcar Fracture: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Calcar Fracture: Absent | 95 | 93
  Week 24: Femoral stem tilt: Present: number analyzed (Participants) | 91 | 88
  Week 24: Femoral stem tilt: Present | 0 | 0
  Week 24: Femoral stem tilt: Absent: number analyzed (Participants) | 91 | 88
  Week 24: Femoral stem tilt: Absent | 12 | 17
  Week 24: Femoral stem tilt: Not applicable: number analyzed (Participants) | 91 | 88
  Week 24: Femoral stem tilt: Not applicable | 79 | 71
  Week 6: Femoral Stem Porous Coating Integrity: Present | 0 | 0
  Week 6: Femoral Stem Porous Coating Integrity: Absent | 75 | 73
  Week 6: Femoral Stem Porous Coating Integrity: Not applicable | 28 | 26
  Week 24: Femoral Stem Porous Coating Integrity: Present: number analyzed (Participants) | 95 | 93
  Week 24: Femoral Stem Porous Coating Integrity: Present | 0 | 0
  Week 24: Femoral Stem Porous Coating Integrity: Absent: number analyzed (Participants) | 95 | 93
  Week 24: Femoral Stem Porous Coating Integrity: Absent | 69 | 67
  Week 24: Femoral Stem Porous Coating Integrity: Not applicable: number analyzed (Participants) | 95 | 93
  Week 24: Femoral Stem Porous Coating Integrity: Not applicable | 26 | 26

13. Secondary Outcome: Number of Participants With Radiographic Outcomes: Femoral Stem Position
Description: Number of participants with radiographic outcome (femoral stem position) were reported. Femoral stem position was assessed as neutral, varus and valgus.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Participants
  Week 6: Neutral | 91 | 82
  Week 6: Varus | 10 | 16
  Week 6: Valgus | 2 | 1
  Week 24: Neutral: number analyzed (Participants) | 95 | 93
  Week 24: Neutral | 83 | 76
  Week 24: Varus: number analyzed (Participants) | 95 | 93
  Week 24: Varus | 10 | 16
  Week 24: Valgus: number analyzed (Participants) | 95 | 93
  Week 24: Valgus | 2 | 1

14. Secondary Outcome: Number of Participants With Radiographic Outcomes: Device/Anatomy Condition
Description: Number of participants with radiographic outcome (device/anatomy condition) were reported. Assessments were reported as intact or not intact.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Participants
  Week 6: Intact | 103 | 99
  Week 6: Non-intact | 0 | 0
  Week 24: Intact: number analyzed (Participants) | 95 | 93
  Week 24: Intact | 95 | 93
  Week 24: Non-intact: number analyzed (Participants) | 95 | 93
  Week 24: Non-intact | 0 | 0

15. Secondary Outcome: Number of Participants With Radiographic Outcomes: Heterotopic Ossification
Description: Number of participants with radiographic outcome (heterotopic ossification) were reported. Ossification is defined as formation of extraskeletal bone in muscle and soft tissues. Heterotopic ossification is the presence of bone in soft tissue where bone normally does not exist. Heterotopic ossification was classified as Class 0, I, II, III and IV where Class 0 indicates "no evidence heterotopic bone formation", Class I indicates "islands of bone within the soft tissue about the hip", Class II indicates "bone spurs from the pelvis or proximal end of the femur, leaving at least a centimeter (cm) between opposing bone surfaces", Class III indicates "bone spurs from the pelvis or proximal end of the femur, reducing the space between opposing bone surfaces to less than 1 cm", and Class IV indicates "apparent bone ankylosis of the hip."
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Participants
  Week 6: Class 0 | 100 | 89
  Week 6: Class I | 2 | 9
  Week 6: Class II | 1 | 0
  Week 6: Class III | 0 | 1
  Week 6: Class IV | 0 | 0
  Week 24: Class 0: number analyzed (Participants) | 95 | 93
  Week 24: Class 0 | 90 | 81
  Week 24: Class I: number analyzed (Participants) | 95 | 93
  Week 24: Class I | 4 | 10
  Week 24: Class II: number analyzed (Participants) | 95 | 93
  Week 24: Class II | 1 | 2
  Week 24: Class III: number analyzed (Participants) | 95 | 93
  Week 24: Class III | 0 | 0
  Week 24: Class IV: number analyzed (Participants) | 95 | 93
  Week 24: Class IV | 0 | 0

16. Secondary Outcome: Radiographic Outcomes: Assessment of Acetabular Cup Version (Hip) and Acetabular Cup Inclination
Description: Radiographic outcome was assessed on acetabular cup version (hip) and acetabular cup inclination and reported in this outcome measure.
Time Frame: Weeks 6 and 24 (post-operative)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 103 | 99
Degrees
  Week 6: Acetabular Cup Version: Hip: number analyzed (Participants) | 101 | 94
  Week 6: Acetabular Cup Version: Hip | 25.2 (2.83) | 25.3 (2.70)
  Week 24: Acetabular Cup Version: Hip: number analyzed (Participants) | 95 | 92
  Week 24: Acetabular Cup Version: Hip | 25.3 (2.72) | 25.2 (2.33)
  Week 6: Acetabular Cup Inclination | 43.9 (3.83) | 43.8 (3.79)
  Week 24: Acetabular Cup Inclination: number analyzed (Participants) | 95 | 93
  Week 24: Acetabular Cup Inclination | 43.8 (3.71) | 43.6 (3.57)

17. Secondary Outcome: Length of Hospital Stay After Index Total Hip Arthroplasty (THA)
Description: Length of hospital stay (in days) after index THA was calculated from date of discharge minus date of surgery.
Time Frame: From operative day (Day 0) to date of discharge (any time from Day 0 to Day 5)
Population: Per protocol population set consisted of all enrolled participants who successfully received planned treatment, who met all inclusion/exclusion criteria, who were seen at least once at post-operative visit, who did not had any protocol deviation which were prospectively determined to potentially had influence on scientific validity of data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 109 | 109
Days | 0.8 (0.75) | 0.7 (0.65)

18. Secondary Outcome: Number of Participants With Re-hospitalization During the Study
Description: Number of participants with re-hospitalizations during the study was reported.
Time Frame: Day 0 (operative day) to Day 90 (post-operative)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 109 | 109
Participants | 0 | 1

19. Secondary Outcome: Number of Participants With Narcotic Pain Medication Usage
Description: Number of participants who received any narcotic pain medication to manage study hip pain was reported.
Time Frame: From post operation (Day 0) to Week 24
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 109 | 109
Participants | 99 | 100

20. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Number of participants who experienced post-operative complication was reported.
Time Frame: Day 0 (operative day) up to Week 24
Population: The safety population set consisted of all participants in the enrolled population set for whom treatment was attempted, according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
Number analyzed (Participants) | 117 | 111
Participants | 13 | 10

ADVERSE EVENTS:
Time Frame: From Baseline (Day 0) up to end of study (up to 31 months)
Description: The safety population set consisted of all enrolled participants who signed the informed consent document and attempted treatment according to the actual treatment received.
Arm/Group | Arm 1: KINCISE | Arm 2: MALLET
All-Cause Mortality (participants affected / at risk) | 0/117 | 1/111
Serious Adverse Events (participants affected / at risk) | 0/117 | 3/111
Other Adverse Events (participants affected / at risk) | 21/117 | 8/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: KINCISE (N=117) | Arm 2: MALLET (N=111)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: KINCISE (N=117) | Arm 2: MALLET (N=111)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early due to business decision and not related to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT04191733/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04191733/SAP_001.pdf